CLINICAL TRIAL: NCT06583824
Title: Incidence and Complications Associated with Acquired Swallowing Disorder in the Intensive Care Unit in Extubated or Tracheotomized Patients: a Cohort Study
Brief Title: Incidence and Complications of Post-extubation and Post-tracheostomy Dysphagia in Adult Patients in the Critical Care Unit
Status: Not yet recruiting | Type: Observational
Sponsor: Complejo Hospitalario Universitario de Albacete (Other)
Responsible Party: Principal Investigator, Francisca Calero Yañez, Graduada en Enfermeria, Complejo Hospitalario Universitario de Albacete
Other Study IDs: Chospab
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Complications; Pneumonia; Quality of Lifte; Death; Swallowing Disorder.Other Specified
Keywords: dysphagia; tracheostomy; aspiration; malnutrition; critical care; mechanical ventilation; pneumonia
MeSH Terms: conditions — Pneumonia; Death; Deglutition Disorders; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Acquired Swallowing Disorder in ICU (ICU-ASD), also known as postextubation dysphagia, is a multicausal problem experienced by survivors in intensive care units (ICUs) when the efficiency, safety of swallowing, or both are compromised. These alterations can lead to an increased risk of aspiration, respiratory complications, and malnutrition, potentially resulting in prolonged hospitalization, reduced quality of life, poorer clinical outcomes, and even death.

Despite the clinical and social significance of this disorder, there is limited research addressing it. Existing studies primarily focus on incidence and associated factors, with scant attention to the occurrence of complications, and there is a lack of assessment of the quality of life of these patients. In our context, healthcare professionals are increasingly recognizing the importance of this issue, although the real incidence of ICU-ASD, as well as the frequency of respiratory and nutritional complications, remains unknown. Furthermore, the quality of life of patients with this disorder has not been evaluated thus far.

Objectives:Primary: To analyze the occurrence of respiratory and nutritional complications associated with ICU-ASD in patients intubated for ≥48 hours or tracheotomized in the Intensive Care Unit of the University Hospital Complex of Albacete (ICU CHUA) and identify potential factors related to their occurrence.

Specific: To determine the incidence of ICU-ASD in the polyvalent ICU CHUA, assess the frequency of respiratory complications, evaluate nutritional status, assess quality of life, and determine the mortality of study participants.

Material and Method: Prospective observational cohort study. Setting: Polyvalent ICU CHUA. Participants: Intubated patients for ≥48 hours or tracheotomized, with signed consent. Sampling: Consecutive. Sample size: 414 participants. Demographic/clinical variables. Outcome variables: Occurrence of respiratory complications, nutritional status, quality of life. Instruments: Modified Volume-Viscosity Swallowing Test (mV-VST), Swallowing Quality of Life Questionnaire (SWAL-QoL). Dysphagia detection will occur 24 hours post-extubation and/or 4 days after tracheotomy. Follow-up during hospitalization and post-ICU discharge until the outpatient consultation. Statistical analysis: Absolute and relative frequencies, measures of central tendency and dispersion, significance level of p < 0.05, 95% CI; Bivariate analysis: Checking group homogeneity and hypothesis testing: Chi-square, Student's t-test, U-Mann-Whitney, ANOVA, or Kruskal-Wallis.

DETAILED DESCRIPTION:
Hypothesis: Patients with ICU-Acquired Swallowing Disorder (ICU-ASD) have a higher frequency of respiratory complications and poorer nutritional status compared to patients without dysphagia.

Objectives:

Primary Objective: To analyze the occurrence of respiratory and nutritional complications associated with ICU-Acquired Swallowing Disorder (ICU-ASD) in patients intubated for more than 48 hours or tracheostomized in the multidisciplinary ICU at CHUA, and to explore potential factors related to their occurrence.

Secondary Objectives:

To determine the incidence of ICU-ASD in the multidisciplinary ICU at CHUA. To determine the frequency of respiratory complications in post-extubated and tracheostomized patients in the multidisciplinary ICU at CHUA.

To assess the nutritional status of post-extubated and tracheostomized patients in the multidisciplinary ICU at CHUA.

To evaluate the quality of life with dysphagia in patients who developed ICU-ASD after hospital discharge.

To determine the mortality rate of post-extubated and tracheostomized patients in the ICU at CHUA.

SAMPLE SIZE: Since there is no existing data on complications caused by dysphagia in our unit, we have considered the study by McIntyre et al. (2022), which shows an incidence of pneumonia of 21% in patients with ICU-ASD and 9% in extubated patients without dysphagia (OR=2.51; 95% CI 1.27-4.95). Based on these premises, the sample size was calculated using the Epiinfo® program, estimating a 95% confidence interval (CI), 80% power, and a 1:1 group ratio. We obtain a sample of 360 participants, adding 15% for potential losses, which means an additional 54 patients. The final sample size to be achieved is 414 participants. Participants will be selected through consecutive sampling, meeting inclusion criteria, and always with signed consent after verbal information and delivery of the information sheet. According to statistical data from the CHUA ICU from previous years, achieving this sample will likely take two years.

RECRUITMENT PERIOD: September 2024-September 2026 (2 years) STUDY COMPLETION: Completion of the study until the end of follow-up, death, or withdrawal of informed consent.

VARIABLES AND MEASUREMENT INSTRUMENTS:

Age (difference between date of birth and admission date). Collected from the medical record.

Sex (male/female). As recorded in the medical record. Comorbidities (personal history of disease). Collected from the medical record. Categorized admission diagnosis: cardiovascular, respiratory, gastrointestinal, neurological, trauma, metabolic, hematological, urological, intoxications, and others. These may be later analyzed as two groups: NEUROCRITICAL/NON-NEUROCRITICAL.

Presence of NG tube and number of days. Number and type (Levin®, Flekka®, nasojejunal). Collected from the patient's daily ICU chart.

Endotracheal tube used: number and type (subglottic/non-subglottic). Collected from the vital signs chart.

Tracheostomy: technique used for insertion (PERCUTANEOUS/SURGICAL), cannula number, and type (with cuff/without cuff). Collected from the patient's vital signs chart.

Days of pre-ICU admission (ICU admission date - hospital admission date). Collected from the medical record.

Days of ICU admission (date of transfer to the ward or death - ICU admission date). Collected from the medical record.

Days of post-ICU admission (from transfer to the ward until discharge). Collected from the medical record.

Total hospital stay (day of discharge - day of admission). Collected from the medical record.

Days with invasive mechanical ventilation (IMV). Collected from the ICU vital signs chart.

Days with endotracheal tube (ETT). Collected from the ICU vital signs chart. Days with tracheostomy. Collected from the ICU vital signs chart. Discharge destination (home/healthcare facility). Collected from the medical record, at the time of nursing discharge.

Patient severity in ICU using the Acute Physiology And Chronic Health Evaluation (APACHE) II. Collected from the patient's medical record.

Sequential Organ Failure Assessment (SOFA). Collected from the patient's medical record.

Nutritional parameters:

Body Mass Index (BMI). We will collect weight and height, referring to the baseline state. Weight measurement: when oral feeding begins, the patient will be weighed on a chair or bed scale. Upon transfer to the ward (chair scale). At one month and three months in the post-ICU clinic. Height measurement: the first time it is possible to measure with a stadiometer.

Biochemical parameters: prealbumin, cholesterol, and C-reactive protein (CRP). Collected from the medical record. The week the swallowing test is performed, the day of transfer to the ward, at discharge, and at 30 days in the clinic.

Existence of ICU-ASD determined using the mV-VST13. To perform the test, the patient must have an adequate level of consciousness, RASS 0, and CAM-ICU negative. The test will always be performed before starting oral intake. If positive, indicating ICU-ASD, it will be repeated weekly, in the ward each week while positive. If it remains positive, it will be followed up in the endocrinology clinic, so data from their assessments will be collected.

Respiratory complications:

Respiratory infections. We collect diagnoses of TRACHEOBRONCHITIS and PNEUMONIA described in the medical record. The diagnosis can occur throughout the follow-up, including visits to the health center and emergency services. Record the date from the medical record.

Bronchoaspiration. Described in the medical record as confirmed or suspected. Bronchoaspiration yes/no and the date it occurs.

Reintubation yes/no. Number of times. Collected from the ICU vital signs chart. Hospital readmissions due to swallowing disorder complications. As described in the admission note. Collected from the computerized medical record.

Emergency visits due to swallowing disorder complications. Collected from the computerized medical record.

Quality of life, using the Swallowing Quality of Life Questionnaire for adults (SWAL-QoL). The SWAL-QoL consists of 44 items distributed in 11 domains: meal duration, desire to eat, food selection, communication, burden, fear, social role, mental health, fatigue, and sleep. It is easy to apply and provides information on self-perception of quality of life. It assesses the impact of dysphagia on the patient, symptoms, how dysphagia affects food choices, the social impact of dysphagia, among others. Each item is rated from 1 to 5 (1 represents the worst state and 5 represents the most favorable state) and is grouped into 10 scales that are evaluated independently (with 0% being the least favorable and 100% the most favorable). Lower scores are associated with poorer quality of life.

Death yes/no. If it occurs from inclusion in the study until its completion. If it occurs, the date of death will be recorded. Collected from the medical record.

Nutritional adaptation. Prescribed diet (type of hospital diet or enteral nutrition) and route of administration: oral, NG tube, or percutaneous endoscopic gastrostomy (PEG).

An ad hoc data collection form has been developed, where all study variables will be recorded on a sheet for each participant. Data will be safeguarded to preserve participants' privacy and confidentiality, and a database will be created for subsequent analysis.

Data Collection

After receiving approval from the Research Ethics Committee for Medicines (CEIm) of the Albacete Health Area, as well as authorization from the department head and ICU supervisor at CHUA, and once the suitability of the facilities has been verified, data collection will begin for those patients who meet the inclusion criteria and sign the informed consent, after having received verbal information. All participants will undergo dysphagia assessment using the mV-VST, and the recording of variables in the specially designed data collection notebook will commence.

The mV-VST is based on testing three textures: nectar, pudding, and liquid, prepared with mineral water and a thickener. In this study, the thickener currently available in the unit will be used, and the staff will be properly trained in its use. The test begins with the nectar texture, gradually increasing the volumes to 5, 10, and 15 ml, which are deposited consecutively into the mouth using a wide-cone 50 ml syringe. These textures will be colored with blue food coloring to better visualize possible pulmonary aspirations, distinguishing them from normal secretions, which is especially important in tracheotomized patients.

For each texture, the following safety criteria must be met: (1) presence of a cough, (2) desaturation greater than 3%, (3) changes in voice tone (not applicable for tracheotomized patients), and (4) presence of esophageal residue, asking the patient if they feel they haven't swallowed everything. If there is no alteration in these parameters with the nectar texture, the same process will be followed with the pudding and liquid textures in that order.

Liquid is the last viscosity tested because ICU patients have great difficulty swallowing liquids. After six intakes at the end of the mV-VST, fatigue may worsen dysphagia due to ICU-AW (ICU-acquired weakness), making the risk of aspiration when ingesting liquids more evident. Unlike the original V-VST, which considers the presence of pharyngeal residue as a measure of efficacy, we evaluate it as a safety parameter, as ICU patients with dysphagia are more likely to experience pulmonary aspiration of pharyngeal residue due to reduced strength to clear it back to the mouth. Dysphagia and aspiration risk will only be ruled out for patients who show safe swallowing for all tested volumes and viscosities in the mV-VST. If any safety parameter is altered, the evaluation will be interrupted, diagnosing ICU-ASD and aspiration risk. A test will be considered POSITIVE, and ICU-ASD will be diagnosed when a YES appears in the corresponding box on our data collection sheet, meaning that the patient has not tolerated that texture because a safety parameter has been affected (e.g., presence of cough, desaturation >3%, change in voice tone, or appearance of pharyngeal residue).

To perform the mV-VST, post-extubated patients must have been intubated for ≥48 hours, and the test will be conducted 24 hours after extubation. For tracheotomized patients, we will wait four days after stoma creation to conduct the test, and these patients must be disconnected from invasive mechanical ventilation for at least 6 hours a day.

Patients must be awake, conscious, and cooperative, with a RASS = 0 and a negative CAM-ICU. During the procedure, the patient will remain seated in bed (at least 45°) or in a chair and will be monitored throughout. For tracheostomized patients, the test will be performed with the cuff deflated and, for those who can tolerate it, with a speaking valve.

Patient identification will be done using a consecutive inclusion number in the study, respecting data confidentiality.

The weight recorded at admission will be the one reported by the patient or family (considering the impossibility of weighing patients due to clinical instability upon ICU admission). After extubation, weight will be recorded either from the bed scale or chair scale (depending on the patient's condition). Height will be recorded when it is possible to measure the patient using a stadiometer (same brand and model available throughout CHUA).

The patient will follow the usual practice in both the ICU, hospitalization ward, and post-ICU clinic. The occurrence of outcome variables will be monitored, including respiratory complications and readmissions, as well as the nutritional status being evaluated.

Based on the mV-VST result, the patient's diet will be adapted, or if oral feeding is impossible, it will be decided whether to administer enteral nutrition via NGT (nasogastric tube) or PEG (percutaneous endoscopic gastrostomy), which will be recorded in the clinical history, and the investigators will document.

During hospitalization and after ICU discharge, the patient will be followed up, recording the results of dysphagia evaluations performed (if continued to be necessary), noting anthropometric and biochemical parameters, and monitoring the occurrence of outcome variables.

After hospital discharge, patients will be monitored through computerized clinical history, looking for new admissions due to complications, as well as visits to their health center or emergency department.

Patients are usually scheduled for post-ICU follow-up visits at 30 and 90 days after hospital discharge. During these visits, the mV-VST will be reevaluated if necessary, and at the 90-day visit, the perceived quality of life will be assessed using the Swallowing Quality of Life Questionnaire for the adult population (SWAL-QoL).

ELIGIBILITY:
Inclusion Criteria:

Patients aged ≥ 18 years, requiring intubation for ≥ 48 hours and/or subsequent tracheostomy, with an adequate level of consciousness to perform the dysphagia diagnostic test, and who have signed the consent form.

Exclusion Criteria:

Previous tracheostomy, prior diagnosis of dysphagia, neurodegenerative disease, or a history of stroke (CVA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the multidisciplinary ICU at CHUA who require intubation or tracheostomy during their stay. CHUA is a tertiary-level hospital with approximately 700 beds, and it is part of the Integrated Healthcare Management of Albacete under the Health Service of Castilla-La Mancha (SESCAM). The multidisciplinary Intensive Care Unit is located on the second floor, central area, of the General Hospital. It is a general (multidisciplinary) unit that manages all critical pathologies (along with other critical care units in the Hospital Complex) except for pediatric cases. The multidisciplinary ICU currently has 18 functional beds, and the majority of admissions are due to medical conditions.
Sampling Method: Non-Probability Sample
Enrollment: 414 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory Complications | This outcome variable may appear from the completion of the mV-VST until the end of participation 90 days after hospital discharge.
  Pneumonia: when a new pulmonary infiltrate or progression appears on the chest x-ray, or cavitation or consolidation, associated with at least 2 of the following criteria: temperature > 38oC, leukocyte count > 12,000/mm3 or leukocytopenia < 4,000/mm3, purulent orotracheal secretion or change in the characteristic of sputum, increased secretions and need for greater suction, new respiratory sounds or rales, worsening oxygenation.
  tracheobronchitis: clinical syndrome similar to pneumonia that must meet at least 2 of the aforementioned criteria, without radiographic infiltrate present.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Macht M, Wimbish T, Bodine C, Moss M. ICU-acquired swallowing disorders. Crit Care Med. 2013 Oct;41(10):2396-405. doi: 10.1097/CCM.0b013e31829caf33. PMID 23939361
- [Background] McInytre M, Doeltgen S, Shao C, Chimunda T. The incidence and clinical outcomes of postextubation dysphagia in a regional critical care setting. Aust Crit Care. 2022 Mar;35(2):107-112. doi: 10.1016/j.aucc.2021.03.008. Epub 2021 May 24. PMID 34034939
- [Background] Schefold JC, Berger D, Zurcher P, Lensch M, Perren A, Jakob SM, Parviainen I, Takala J. Dysphagia in Mechanically Ventilated ICU Patients (DYnAMICS): A Prospective Observational Trial. Crit Care Med. 2017 Dec;45(12):2061-2069. doi: 10.1097/CCM.0000000000002765. PMID 29023260
- [Background] Martinez de Lagran Zurbano I, Laguna LB, Soria CV, Guisasola CP, Marcos-Neira P. Utility of the modified Volume-Viscosity Swallow Test for bedside screening of dysphagia in critically ill patients. Clin Nutr ESPEN. 2023 Feb;53:214-223. doi: 10.1016/j.clnesp.2022.12.021. Epub 2022 Dec 23. PMID 36657916
- [Background] Zaldibar-Barinaga MB, Miranda-Artieda M, Zaldibar-Barinaga A, Pinedo-Otaola S, Erazo-Presser P, Tejada-Ezquerro P. Versión española del Swallowing Quality of Life Questionnaire: fase inicial de adaptación transcultural. Rehabilitación. 2013;47(3):136-40.
- [Background] McIntyre M, Doeltgen S, Dalton N, Koppa M, Chimunda T. Post-extubation dysphagia incidence in critically ill patients: A systematic review and meta-analysis. Aust Crit Care. 2021 Jan;34(1):67-75. doi: 10.1016/j.aucc.2020.05.008. Epub 2020 Jul 29. PMID 32739246
- [Background] Skoretz SA, Flowers HL, Martino R. The incidence of dysphagia following endotracheal intubation: a systematic review. Chest. 2010 Mar;137(3):665-73. doi: 10.1378/chest.09-1823. PMID 20202948